CLINICAL TRIAL: NCT03623919
Title: FallSensing Multiplayer Games for Fall Risk Prevention in Senior Care Centers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Escola Superior de Tecnologia da Saúde de Coimbra (Other)
Collaborators: Sensing Future Technologies (Other); Fraunhofer Portugal Research Center for Assistive Information and Communication Solutions (Other)
Responsible Party: Principal Investigator, Anabela Correia Martins, Senior Lecturer Physiotherapy Dept., Escola Superior de Tecnologia da Saúde de Coimbra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Accidental Fall

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise group (Experimental): Group games, including two teams of seniors aged 50 years or older. The FallSensing games software include 3 mini-games to be played by two teams with up to 3 players each will compete against each other alternately.
  The players will perform an initial evaluation with FallSensing screening tool, 16 sessions of group games (2 times a week/8weeks) with FallSensing multiplayer games and a final evaluation also with FallSensing screening tool.
  Both initial and final evaluation include six functional tests (Grip Strength, Timed Up and Go, 30 seconds Sit-to-Stand, Step test, 4 Stage Balance test "modified" and 10 meters Walking Speed) and a questionnaire concerning self-efficacy for Exercise.
  Interventions: Other: FallSensing multiplayer games

INTERVENTIONS:
Other: FallSensing multiplayer games — FallSensing multiplayer games is a technological solution based on an interactive (exer)game.
  Players will wear a strap on the lower limbs contaning an inertial sensor. This device enables movement identification on the characterization in real time, triggering actions in the game.
  The exercise games are based on a validated fall prevention exercise plan - the Otago Exercise Programme. The exercises were designed to promote mobility and improve muscle strength and balance.

SUMMARY:
Fall prevention programs should include strength and balance training, home hazard assessment and intervention, vision assessment and referral and also medication review with modification/withdrawal. Evidence exists that a tailored exercise program can reduce falls by as much as 54%.

The FallSensing games software include 3 mini-games to be played by two teams with up to 3 players each will compete against each other alternately.

The players will perform an initial evaluation with FallSensing screening tool, 16 sessions of group games (2 times a week/8weeks) with FallSensing multiplayer games and a final evaluation also with FallSensing screening tool.

Both initial and final evaluation include six functional tests (Grip Strength, Timed Up and Go, 30 seconds Sit-to-Stand, Step test, 4 Stage Balance test "modified" and 10 meters Walking Speed) and a questionnaire concerning self-efficacy for Exercise.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 50 years or over;
* Community-dweller;
* independent to be standing and walking, with or without walking aids;
* interest to participate in the study.

Exclusion Criteria:

* individuals with severe sensorial impairments (deafness or blindness)
* individuals with cognitive impairments which precludes the ability to comprehend the questionnaire, functional tests and exercises included in the protocol.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
30 seconds Sit-to-Stand | Change from baseline 30 seconds Sit-to-Stand score up to 8 weeks
  number of stands
4 Stage Balance Test "Modified" | Change from baseline 4 Stage Balance Test "Modified" score up to 8 weeks
  last position accomplished
Self-efficacy for Exercise | Change from baseline Self-efficacy for exercise score up to 8 weeks
  Score 5 to 20 points (the higher the score, the better Self-efficacy)

SECONDARY OUTCOMES:
Timed Up and Go | Outset and up to 8 weeks
  seconds
Grip Strength | Outset and up to 8 weeks
  Kilogram-force
Step Test | Outset and up to 8 weeks
  number of steps
10 meters Walking Speed | Outset and up to 8 weeks
  meters per second

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Tecnologia da Saúde de Coimbra, Coimbra, Portugal